CLINICAL TRIAL: NCT05047549
Title: Community-based RSV Surveillance in Infant Mortality: Minimally Invasive Tissue Sampling Study in Karachi, Pakistan
Acronym: RSV-MITS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: RTI International (Other); Bill and Melinda Gates Foundation (Other); Yale University (Other)
Responsible Party: Principal Investigator, Dr Abdul Momin Kazi, Assistant Professor, Aga Khan University
Other Study IDs: 2020-3675-10613
Record Dates: First submitted 2020-11-23; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Syncytial Virus (RSV); Infant Death; Community-Acquired Infections
Keywords: respiratory syncytial virus; infant mortality; minimally invasive tissue sampling
MeSH Terms: conditions — Infant Death; Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to assess the burden of respiratory syncytial virus on infant mortality in Pakistan, nasopharyngeal swab sampling and minimally invasive tissue sampling (MITS) will be conducted on deceased infants under 6 months of age. The specimens will be analysed by the microbiology and histopathology labs at Aga Khan University, Karachi, Pakistan. Verbal consent will be obtained from parents of deceased infants, and a cause of death lab report and grief counseling services will be offered to enrolled parents who gave consent for specimen collection. The study is funded by Bill & Melinda Gates Foundation in affiliation with Research Triangle Institute (RTI) MITS Surveillance Alliance.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is a respiratory pathogen with potentially high disease burden in Lower middle income country (LMIC). This pathogen is a potential target for maternal immunization strategies to prevent disease and early death in young infants. Majority of current studies estimate the burden of disease in terms of facility-based (e.g. hospital) deaths. There is a knowledge gap regarding the proportion of community-based deaths due to RSV. There are many challenges to generating evidence for the burden of RSV, such as lack of resources for hospital and community surveillance and diagnostics, and difficulty in obtaining specimens.

Parent study: In January 2018, the Community-based Infant RSV Mortality Study was initiated in collaboration with Emory University, funded by the Bill and Melinda Gates Foundation. Following a formative phase involving interviews with community stakeholders, in August 2018 a pilot surveillance stage was initiated, in which upon receiving death alerts from key community partners about the recent death of an infant (<6 months) in the 4 catchment areas of Karachi, a team of nurses and health workers mobilize to identify and approach the household of the infant's primary caregivers. Upon obtaining verbal consent from the parents, the nurse obtains nasopharyngeal specimens from the left and right nostrils of the recently deceased infant. These specimens are tested for respiratory syncytial virus and Bordetella pertussis through real-time Polymerase chain reaction (PCR) testing, and lab results are reported to the parents along with verbal autopsy findings in a cause of death consultation. Enrolled bereaved parents are also offered grief support home visits and grief counseling services by the community health workers and study psychologist. The surveillance phase continued from August 2018 to March 2020, when specimen collection was paused due to coronavirus disease of 2019 (COVID-19) distancing measures. In 20 months, 490 nasopharyngeal specimens were collected out of 713 households approached upon death alerts. Of these 490, 14 tested positive for RSV and 1 positive for pertussis. Following a training on disinfection, personal protective equipment (PPE) protocols, distancing measures, as well as a study-specific training on mental health, communication, and counseling skills June-July 2020, surveillance and specimen collection is planned to resume from August 2020.

Proposal for current study: While nasopharyngeal swab sampling with PCR testing is the gold standard for detection of RSV, little is understood about lung morphology in relation to upper respiratory tract infections in neonate and infant mortality. The objective of this study is to assess and analyze the burden and determinants of RSV mortality in infants in 2 peri-urban areas of Karachi Pakistan and to provide a cause of death consultation for the families of the recently deceased infants under 6 months of age in the catchment areas.

The RSV-MITS Study will be merged with the ongoing parent study of Community-based Infant RSV Mortality. With the additional procedure and analysis of minimally invasive tissue sampling (MITS) of the lungs/thorax, we aim to examine lung morphology through microbiology and histology specimens. Designated staff (nurses) will require additional MITS training, and the nasopharyngeal swab specimens and lung/thorax MITS specimens will be collected in the designated study ambulance parked near the household or transported to the closest partner hospital. The target sample size is 150 lung/thorax MITS and nasopharyngeal specimens from deceased infants under 6 months of age; stillbirths and miscarriages excluded. This study will be conducted in 2 Health and Demographic Surveillance System (HDSS) catchment areas: Bhains Colony and Ali Akbar Shah Goth. The MITS Study is funded by the MITS Surveillance Alliance.

ELIGIBILITY:
Inclusion Criteria:

* Parents, caregivers of deceased infants (under 6 months of age)
* Residing in one of 2 catchment areas in Karachi, enrolled in Demographic Surveillance System
* Have given informed verbal consent for collection of nasopharyngeal specimen AND lung/thorax tissue sampling

Exclusion Criteria:

* Miscarriages (under 28 gestational weeks)
* Known stillbirths
* Guest/visiting families in the area that will not be participating in verbal autopsy after infant death

Ages: 1 Minute to 6 Months | Sex: All
Age Groups: Child
Study Population: Deceased neonates and infants (under 6 months of age) born and died within specified catchment areas
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
RSV nasopharyngeal swab | 2 months
  A special swab will be use to take a sample from the nose or throat and Reverse transcription-Polymerase chain reaction (RT-PCR) will be done to understand the burden of disease in deceased children under 6 months of age from a real time community setting.
RSV lung/thorax microbiology | 2 months
  lung fluid will be aspirated and Reverse transcription-Polymerase chain reaction (RT-PCR) will be done to assess the burden of RSV in deceased infants under 6 months of age.
RSV lung/thorax histopathology | 2 months
  Minimally invasive tissue sampling (MITS) will be performed to obtain lung tissue specimens Tissues will be examined through histopathology. Through the sample collection we will understand the burden of RSV among deceased infants, as well as cause of death due to upper respiratory tract infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan